CLINICAL TRIAL: NCT04713007
Title: Improving Quality of Life for Colon Cancer Patients and Their Caregivers
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hawaii (Other)
Collaborators: Alliance for Clinical Trials in Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Cassel 2020-2
Record Dates: First submitted 2020-12-29; First posted 2021-01-19 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Experimental): Supportive Care Materials and Resources
  Interventions: Behavioral: Quality of Life Supportive Resources
- Group A (Experimental): Ted Talks/Educational videos
  Interventions: Behavioral: Quality of Life Ted Talks

INTERVENTIONS:
Behavioral: Quality of Life Ted Talks — There will be 9 training modules released weekly on the tablet. A survey will be required at baseline, each of the 9 weeks and at 3 months.
  Arms: Group A
Behavioral: Quality of Life Supportive Resources — The tablet will be preloaded with cancer information and supportive care resources from the National Cancer Institute. A survey will be required at baseline, each of the 9 weeks and at 3 months.
  Arms: Group 1

SUMMARY:
By joining this study, participants, including patients and their caregivers, will be provided useful information about colon cancer that may help alleviate anxiety surrounding treatment, improve communications with the medical team, and identify practical ways to support each other. Participating in this study will have no impact on your cancer care that participants receive from your provider. It is expected that the resources provided to participants and participants caregiver will help improve participants overall care. The study team will provide computer tablets for patients and their caregivers to use as part of the study to access information about colon cancer and how to help manage participants therapeutic care. The study team will check-in each week to provide assistance with the use of the tablets and ask the patient and their caregiver, to complete an assessment survey.

As part of the surveys the study team will collect participants full name, address and phone number and some basic information about participants (e.g., age, gender and race). The study team will also collect some personal or medical information, including the stage of colon cancer and treatment received (if the participant) or your relationship to the patient if participants caregiver. The study team will also collect some information on your emotional health and views about the medical care that has been provided to date from the questionnaire. All this information will be held confidential and not forwarded to anyone outside of the study personnel. There are no activities required, except that the study team will encourage caregivers and patients to discuss and use the information provided in computer tablets to enhance their cancer care. Whether or not the participants use this information will not affect their ability to receive high-quality care from their providers.

There is a slight burden of responding to the survey questions used to help us understand the useful features of this program. For this reason, the investigator has included small incentives to support the time and effort needed to complete these survey assessments. The study team hopes that this study, one of the first of its kind, will help identify the resources and methods that can be used to help patients and caregivers have a better understanding of their cancer care and provide resources that they can use to enhance the effectiveness of their therapy.

ELIGIBILITY:
Inclusion Criteria: Patient

* Colon Cancer patients must live in Honolulu County and must identify a patient caregiver
* Patients must have newly diagnosed stage II-III colon cancer and be < 60 days from surgical treatment at the time of registration.
* Adults over age 18
* Adequate understanding of English language and must be able to read and write English
* Must be able to provide informed consent

Exclusion Criteria: Patient

-Patients who are > 60 days from surgical treatment will be ineligible

Inclusion Criteria: Caregiver

* Must live in Honolulu County
* Must either be an adult family member of a colon cancer patient or a patient identified caregiver
* Adults over age 18
* Adequate understanding of English language and must be able to read and write English
* Must be able to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-06-03 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Quality of Life Scores | change from baseline to 3 months
  Compare QOL scores of patients using the EORTC QLQ-C30 instrument at post randomization between intervention and control arm
Quality of Life Scores | change from baseline to 3 months
  Compare QOL scores of caregivers using the CQOLC instrument at post randomization between intervention and control arm
Perception of Care Coordination Participant | change from baseline to 3 months
  Care coordination will be measured using our developed care coordination instruments (CCI), a 29 item, self-reported, multiple choice survey questionnaire
Perception of Care Coordination Caregiver | change from baseline to 3 months
  Care coordination will be measured using our developed care coordination instruments (CCICG), a 29 item, self-reported, multiple choice survey questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Kevin D Cassel, Dr. PH, Principal Investigator — University of Hawaii Cancer Research Center
Locations (4):
- United States (4):
  - Hawaii Cancer Care Inc, Honolulu, Hawaii
  - Hawaii Pacific Health, Honolulu, Hawaii
  - The Queens Medical Center, Honolulu, Hawaii
  - Adventist Health Castle, Kailua, Hawaii

IPD SHARING:
Plan to Share IPD: No